CLINICAL TRIAL: NCT04589793
Title: COaching Lifestyle Intervention for FErtility
Acronym: COLIFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Maritta Poyhonen-Alho, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYH2020338
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Life Style; Fertility Disorders
Keywords: Infertility; Life Style; Physical activity; Diet; Sleep and stress; Intervention; Obesity
MeSH Terms: conditions — Infertility; Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Conventional treatment
- Intervention (Active Comparator): Motivational interview
  Interventions: Behavioral: Life Style

INTERVENTIONS:
Behavioral: Life Style — Life Style intervention including physical activity, diet, sleep and stress
  Arms: Intervention

SUMMARY:
In Finland, every third woman is overweight (BMI>25) and 11,5% obese (BMI>30). Cohort and national studies reveal that 46% of fertile-aged men have BMI≥25 and 20% BMI≥30. Overweight has negative impact on both female and male fertility and weakens markedly the results of infertility treatments. In this study, 780 infertile couples will be randomized to control group (conventional infertility treatment) and lifestyle intervention arm undergoing 4 sessions of video-mediated motivational interview, anthropometric measurements, laboratory tests and epigenetic samples. Economic evaluation of the intervention will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* infertility
* BMI 27-34.9 kg/m2

Exclusion Criteria:

* no mobile device available
* evident sperm defect or ovarian tube block
* hinder for fluent treatment schedule due to the subjec´s obstacle (inadequate language skills, major time table problems)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1560 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Behavior change | 6 months
  score from 1 to 4: (smoking + daily vegetable, fruit and berry use >500g + BMI 19-27 + 150 min of moderate exercise/week) No=0, Yes=1 measured at the beginning, at 3 and 6 months
Live birth rate | 3 years
  Number of live children born
Weight change | 6 months
  weight in kg measured without shoes and with light clothing at the beginning, at 3 and 6 months

SECONDARY OUTCOMES:
Infertility treatments, number | 3 years
  Number of infertility treatments needed for a live birth
Infertility treatments, mode | 3 years
  Mode of infertility treatments needed for a live birth (including ovulation induction, insemination, IVF, ICSI)
Miscarriage rate | 3 years
  Number of miscarriages
Height | 0 months
  Measured without shoes (cm)
Weight | 0 months
  Measured without shoes and with light clothing (kg)
Weight | 3 months
  Measured without shoes and with light clothing (kg)
Weight | 6 months
  Measured without shoes and with light clothing (kg)
Body mass index | 0 months
  Weight in kilograms divided by the square of height in meters
Body mass index | 3 months
  Weight in kilograms divided by the square of height in meters
Body mass index | 6 months
  Weight in kilograms divided by the square of height in meters
Body composition | 0 months
  Bioimpedance method
Body composition | 3 months
  Bioimpedance method
Body composition | 6 months
  Bioimpedance method
Waist circumference | 0 months
  measured at midpoint between the lower margin of the last palpable rib and the top of the iliac crest (cm)
Waist circumference | 3 months
  measured at midpoint between the lower margin of the last palpable rib and the top of the iliac crest (cm)
Waist circumference | 6 months
  measured at midpoint between the lower margin of the last palpable rib and the top of the iliac crest (cm)
Self-reported physical activity | 0 months
  Minutes per week, International Physical Activity Questionnaire - Short Form
Self-reported physical activity | 6 months
  Minutes per week, International Physical Activity Questionnaire - Short Form
Physical activity | 0 months
  Amount of weekly physical activity, data from Oura ring 3-dimensional accelerometer
Physical activity | 3 months
  Amount of weekly physical activity, data from Oura ring 3-dimensional accelerometer
Physical activity | 6 months
  Amount of weekly physical activity, data from Oura ring 3-dimensional accelerometer
Maximal oxygen uptake | 0 months
  Functional aerobic capacity prediction model (N-Ex BMI) by Johnson et al 1990
Maximal oxygen uptake | 3 months
  Functional aerobic capacity prediction model (N-Ex BMI) by Johnson et al 1990
Maximal oxygen uptake | 6 months
  Functional aerobic capacity prediction model (N-Ex BMI) by Johnson et al 1990
Dietary content | 0 months
  FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a)
Dietary content | 6 months
  FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a)
Dietary patterns | 0 months
  FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a)
Dietary patterns | 6 months
  FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a)
Folate | 0 months
  Plasma folate concentration
Folate | 6 months
  Plasma folate concentration
Vitamin-D | 0 months
  Plasma vitamin-D concentration
Vitamin-D | 6 months
  Plasma vitamin-D concentration
Zinc | 0 months
  Plasma zinc concentration
Zinc | 6 months
  Plasma zinc concentration
Carbohydrates | 0 months
  Amount of daily carbohydrates in diet , FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Carbohydrates | 6 months
  Amount of daily carbohydrates in diet, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Protein | 0 months
  Amount of daily proteins in diet, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Protein | 6 months
  Amount of daily proteins in diet, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Alcohol | 0 months
  Alcohol consumption per week, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Alcohol | 6 months
  Alcohol consumption per week, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
n-3 fatty acids | 0 months
  Amount of daily n-3 fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
n-3 fatty acids | 6 months
  Amount of daily n-3 fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
n-6 fatty acids | 0 months
  Amount of daily n-6 fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
n-6 fatty acids | 6 months
  Amount of daily n-6 fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Saturated fatty acids | 0 months
  Amount of daily saturated fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Saturated fatty acids | 6 months
  Amount of daily saturated fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Monounsaturated fatty acids | 0 months
  Amount of daily monounsaturated fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Monounsaturated fatty acids | 6 months
  Amount of daily monounsaturated fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Polyunsaturated fatty acids | 0 months
  Amount of daily polyunsaturated fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Polyunsaturated fatty acids | 6 months
  Amount of daily polyunsaturated fatty acids, FinTerveys dietary questionnaire (https://thl.fi/documents/189940/4779595/FT17_FFQ_ENG_paino.pdf/4a2ef46b-272e-4bb4-827c-e1cb1314f09a
Sleep | 0 months
  Quality of sleep, Basic Nordic Sleep Questionnaire (BNSQ)
Sleep | 6 months
  Quality of sleep, Basic Nordic Sleep Questionnaire (BNSQ)
Sleep, measured | 0 months
  Quality, sleep disruptions, total sleep duration registered by Oura ring application
Sleep, measured | 3 months
  Quality, sleep disruptions, total sleep duration registered by Oura ring application
Sleep, measured | 6 months
  Quality, sleep disruptions, total sleep duration registered by Oura ring application
Stress recovery | 0 months
  Night-time heart rate variability regisered by Oura ring application
Stress recovery | 3 months
  Night-time heart rate variability registered by Oura ring application
Stress recovery | 6 months
  Night-time heart rate variability registered by Oura ring application
Anxiety and depression | 0 months
  Hospital Anxiety and Depression Scale (HADS)
Anxiety and depression | 3 months
  Hospital Anxiety and Depression Scale (HADS)
Anxiety and depression | 6 months
  Hospital Anxiety and Depression Scale (HADS)
Fertility quality of life | 0 months
  FertiQoL International Questionnaire
Fertility quality of life | 6 months
  FertiQoL International Questionnaire
Depression | 0 months
  Edinburgh Postnatal Depression Scale (EPDS) Questionnaire
Depression | 6 months
  Edinburgh Postnatal Depression Scale (EPDS) Questionnaire
Self-determined motivation for physical activity | 0 months
  Behavioral Regulations for Exercise Questionnaire (BREQ-3, Markland, D. & Tobin, 2004). Includes the subscales: Amotivation, External regulation, Introjected regulation, Identified regulation, Integrated regulation, Intrinsic regulation.
Self-determined motivation for physical activity | 6 months
  Behavioral Regulations for Exercise Questionnaire (BREQ-3, Markland, D. & Tobin, 2004). Includes the subscales: Amotivation, External regulation, Introjected regulation, Identified regulation, Integrated regulation, Intrinsic regulation
Intention and action planning for physical activity; Intention to increase physical activity | 0 months
  Three (adapted) items from the Health Action Process Approach Questionnaire, (Schwarzer R. Modeling health behaviour change: how to predict and modify the adoption and maintenance of health behaviors. Appl Psychol, 2008; 57:1-29)
Intention and action planning for physical activity; Intention to increase physical activity | 6 months
  Three (adapted) items from the Health Action Process Approach Questionnaire (Schwarzer R. Modeling health behaviour change: how to predict and modify the adoption and maintenance of health behaviors. Appl Psychol, 2008; 57:1-29)
Self-efficacy for physical activity | 0 months
  18-item scale developed by Albert Bandura (Bandura A. 2006). Guide for constructing self-efficacy scales. In: Pajares F, Urdan T (eds)Self-efficacy beliefs of adolescents. Information Age, Charlotte, pp 307-337)
Self-efficacy for physical activity | 6 months
  18-item scale developed by Albert Bandura (Bandura A. 2006). Guide for constructing self-efficacy scales. In: Pajares F, Urdan T (eds)Self-efficacy beliefs of adolescents. Information Age, Charlotte, pp 307-337)
Pregnancy complications | 3 years
  Number of pregnancy complications (gestational diabetes, pre-eclampsia, hypertension, fetal growth disorders, preterm birth)
Delivery complications | 3 years
  Number of delivery complications (cesarean section, assisted vaginal delivery, hemorrhage)
Neonatal outcome | 3 years
  Birth weight, cord pH, Apgar score
Body composition of the newborn | At birth
  Bioimpedance method
Growth of the child | Up to 16 years of age
  From the records of the national child care centers and schools
Sperm epigenetic profile | 0 months
  Determination of heritable phenotype
Sperm epigenetic profile | 6 months
  Determination of heritable phenotype
Transcriptome | 0 months
  RNA-sequencing
Transcriptome | 6 months
  RNA-sequencing
Sperm oxidative stress | 0 months
  the Male infertility Oxidative System test (MiOXSYS)
Sperm oxidative stress | 6 months
  the Male infertility Oxidative System test (MiOXSYS)
A cost-utility of the intervention | 3 years
  analysis based on WHOQOL-BREF Questionnaire and FertiQoL, relating the quality-adjusted life years (QALYS) to the costs of the intervention
QALY baseline | 0 months
  WHOQOL-BREF Questionnaire and FertiQoL International Questionnaire
QALY end point | 6 months
  WHOQOL-BREF Questionnaire and FertiQoL International Questionnaire
Cost-effectiveness | 3 years
  ICER
Static postural balance | 0 months
  Absolute reach distance measured on balance board, cm (FTC Functional training Company GmbH, AM Haag 10 D-82166 Gräfelfing Germany)
Static postural balance | 1st trimester of pregnancy
  Absolute reach distance measured on balance board, cm (FTC Functional training Company GmbH, AM Haag 10 D-82166 Gräfelfing Germany)
Static postural balance | 2nd trimester of pregnancy
  Absolute reach distance measured on balance board, cm (FTC Functional training Company GmbH, AM Haag 10 D-82166 Gräfelfing Germany)
Static postural balance | 3rd trimester of pregnancy
  Absolute reach distance measured on balance board, cm (FTC Functional training Company GmbH, AM Haag 10 D-82166 Gräfelfing Germany)
Static postural balance | 3 months postpartum
  Absolute reach distance measured on balance board, cm (FTC Functional training Company GmbH, AM Haag 10 D-82166 Gräfelfing Germany)
Perception of stress | 0 months
  Perceived Stress Scale by Sheldon Cohen
Perception of stress | 3 months
  Perceived Stress Scale by Sheldon Cohen
Perception of stress | 6 months
  Perceived Stress Scale by Sheldon Cohen
Personality dimensions | 0 months
  The Big Five Personality Test
Personality dimensions | 6 months
  The Big Five Personality Test

CONTACTS AND LOCATIONS:
Overall Officials: Juha Tapanainen, professor, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No
According to request and after consideration of the study group